CLINICAL TRIAL: NCT02167672
Title: What Would it Take to Reduce the Proportion of Women Who Have a Hysterectomy Via an Open Abdominal Approach in Australia?
Brief Title: Barriers for the Uptake of LaparoScopic Hysterectomy
Acronym: LIgHT
Status: Completed | Type: Observational
Sponsor: Queensland Centre for Gynaecological Cancer (Other Government)
Collaborators: Queensland University of Technology (Other)
Responsible Party: Sponsor
Other Study IDs: LIgHT
Record Dates: First submitted 2014-04-16; First posted 2014-06-19 (Estimated); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Hysterectomy
Keywords: total abdominal hysterectomy, total laparoscopic hysterectomy, vaginal hysterectomy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Consumers: Women who have had a Hysterectomy in the previous 2 years
- Doctors: Obstetricians and Gynaecologists

SUMMARY:
Hysterectomy (surgical removal of the uterus) is the most common major gynaecological operation in women in developed countries. In Queensland, 6000 women require a hysterectomy for irregular periods, benign tumours or pelvic pain every year. Surgical approaches to surgical removal of the uterus (womb) include Laparoscopic Hysterectomy (LH), Vaginal Hysterectomy (VH) and Abdominal Hysterectomy through an abdominal incision (AH).

It is widely accepted that LH and VH are less invasive surgical procedures, cause less bleeding, surgical complications and pain and are associated with quicker recovery from surgery than the more invasive AH. In a clinical trial comparing LH and AH we recently demonstrated that LH outperforms AH with regards to cost effectiveness causing less total health-services cost than AH.

Implementation of LH in Queensland could save $9.8 million every year. Despite the evidence for LH and VH, 2600 hysterectomies (43%) are still performed through an open, abdominal incision. In brief, a common but outdated operation is still performed regularly causing not only unnecessary pain, surgical adverse events and longer hospital stay but also increased healthcare costs.

This study will assess reasons why a significant number of gynaecologists and patients prefer AH over LH (Barriers to the uptake of laparoscopic hysterectomy). We will survey specialist gynaecologists as well as patients who have had a hysterectomy for different health reasons. Based on the information from the survey the investigators will develop an intervention to increase the rate of laparoscopic hysterectomies in Queensland and pilot test it.

ELIGIBILITY:
Inclusion Criteria:

* Obstetricians and Gynaecologists or Women who have had a hysterectomy in the previous 2 years

Exclusion Criteria:

* Women who have had a hysterectomy more than 2 years ago
* Women who had a hysterectomy for cancerous conditions

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Members of RANZCOG community sample
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2014-04 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Questionnaire will identify barriers | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Obermair, Study Chair — Queensland Health
Locations (1):
- University of Queensland, Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No